CLINICAL TRIAL: NCT06508034
Title: Probiotics Preventing Immune Checkpoint Inhibitor-Induced Colitis
Brief Title: Probiotics for the Prevention of Immunotherapy Induced Colitis in Patients Receiving Immunotherapy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in funding status
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210304; NCI-2024-05551 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-012363 (Other: Mayo Clinic Institutional Review Board); MC210304 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (VSL#3® 450B) (Experimental): Patients receive VSL#3® 450B (live freeze-dried lactic acid bacteria probiotic) PO QD at least 3 days prior or 1-2 weeks prior to starting standard care or receiving the next cycle of ICIs and then continue for 12 weeks. Patients also undergo stool and blood sample collections on study.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Live Freeze-Dried Lactic Acid Bacteria Probiotic; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo stool and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Dietary Supplement: Live Freeze-Dried Lactic Acid Bacteria Probiotic — Given PO
  Other Names: VSL#3; VSL3
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The clinical trial tests the use of over-the-counter probiotics VSL#3® 450B in patients receiving immunotherapy. Immunotherapy with monoclonal antibodies, helps the body's immune system attack tumor cells, and interferes with the ability of tumor cells to grow and spread. Immunotherapy can also cause an unfortunate side effect of inflammation of the colon and diarrhea, also known as immune checkpoint inhibitor induced colitis. Immune checkpoint inhibitor induced colitis can occur in up to 45% of patients receiving immunotherapy. Taking probiotics VSL#3® 450B may reduce the chances of developing immune checkpoint inhibitor induced colitis in patients receiving immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the incidence of immune checkpoint inhibitors (ICI)-induced colitis (IIC) in patients with solid malignancies receiving over-the-counter multi-strain probiotic blend and ICIs in both cohorts: (1) anti-Cytotoxic T lymphocyte-associated protein-4 (CTLA-4) +/- anti-programmed cell death-1 (PD-1)/programmed cell death-1 ligand 1 (PD-L1), and (2) anti-PD-1/PD-L1 +/- chemo.

SECONDARY OBJECTIVES:

I. To evaluate the safety of multi-strain probiotic blend in cancer patients receiving ICIs.

II. To evaluate the clinical outcomes related to IIC, including the incidence of IIC, hospitalization, treatment delays, and administration of immunosuppressants.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in gut microbiome with ICIs and multi-strain probiotic blend.

II. To evaluate changes in immune response with ICIs and multi-strain probiotic blend.

OUTLINE:

Patients receive VSL#3® 450B (live freeze-dried lactic acid bacteria probiotic) orally (PO) once daily (QD) at least 3 days prior or 1-2 weeks prior to starting standard care ICIs or receiving the next cycle of ICIs and then continue for 12 weeks. Patients also undergo stool and blood sample collections on study.

After completion of study treatment, patients are followed up at 30 days and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Histologically confirmed solid malignancy
* Will be starting on ICIs or have started ≤ 2 cycles of ICIs

  * For cohort 1: Ipilimumab with or without anti-PD-1/PD-L1 including but not limited to pembrolizumab, nivolumab, cemiplimab, atezolizumab, avelumab, or durvalumab
  * For cohort 2: Anti-PD-1/PD-L1 described above with or without chemotherapy
* Absolute neutrophil count (ANC) ≥ 1000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2 x upper limit of normal (ULN)
* Serum glutamic-oxaloacetic transaminase (SGOT) [aspartate transaminase (AST)] ≤ 2 x ULN
* Albumin ≥ 3 g/dL
* Willing and able to provide research stool and blood samples
* Negative serum pregnancy test done ≤ 7 days prior to enrollment, for women of childbearing potential only
* Capable of providing valid informed consent
* Willing to return to enrolling institution for all study visits (blood draws, etc)

Exclusion Criteria:

* Requires prolonged systemic antibiotic therapy for other condition and recent systemic antibiotic within the past 2 weeks
* Fecal microbiota transplant (FMT) within the past 6 months
* FMT with an associated serious adverse event related to the FMT product or procedure
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of over-the-counter probiotics
* Immunocompromised patients including patients known to be HIV positive or those on chronic steroids > 20 mg prednisone a day or prednisone-equivalent Note: Must be off systemic steroids at least 90 days prior to enrollment. However, topical steroids, inhalants or steroid eye drops are permitted
* History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis
* History of chronic diarrhea
* History of celiac disease
* Currently has a colostomy
* Intraabdominal surgery related to gastrointestinal tract within the last 60 days
* Evidence of active, severe colitis
* History of short gut syndrome or motility disorders
* Requires the regular use of medications to manage bowel hypermotility
* Active autoimmune disease that has required systemic treatment in the ≤ 30 days (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) prior to randomization. Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of immune checkpoint inhibitors (ICI)-induced colitis (IIC) with VSL#3 and ICIs | Up to 14 weeks
  Will be evaluated in patients with solid malignancies in 2 cohorts, including 1) anti-CTLA4 ± anti-PD-1/PD-L1, 2) anti-PD-1/PD-L1 ± chemotherapy respectively. Analysis will be performed in all-treated population, defined as any subject enrolled into the study that received at least 3 days of VSL#3 and anti-PD-1/PD-L1. The statistical analyses will be handled in a descriptive manner. Will be estimated by the number of patients who had IIC divided by the total number of evaluable patients. Two-sided 90% exact confidence intervals for the true incidence rate will be calculated according to the approach of Clopper and Pearson.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post treatment
  Will be evaluated by the safety profile of multi-strain probiotic blend in cancer patients receiving ICIs. Analysis will be performed in all-treated population, defined as any subject enrolled into the study that received at least 3 days of VSL#3 and anti-PD-1/PD-L1. The statistical analyses will be handled in a descriptive manner. Descriptive statistics (frequency table) and histogram will be used to summarize toxicity.
Incidence of hospitalization related to IIC | Up to 14 weeks
  Analysis will be performed in all-treated population, defined as any subject enrolled into the study that received at least 3 days of VSL#3 and anti-PD-1/PD-L1. The statistical analyses will be handled in a descriptive manner. Descriptive statistics (frequency table) and histogram will be used to summarize clinical outcomes related to IIC.
Incidence of treatment delays related to IIC | Up to 14 weeks
  Analysis will be performed in all-treated population, defined as any subject enrolled into the study that received at least 3 days of VSL#3 and anti-PD-1/PD-L1. The statistical analyses will be handled in a descriptive manner. Descriptive statistics (frequency table) and histogram will be used to summarize clinical outcomes related to IIC.
Incidence of administration of immunosuppressants related to IIC | Up to 14 weeks
  Analysis will be performed in all-treated population, defined as any subject enrolled into the study that received at least 3 days of VSL#3 and anti-PD-1/PD-L1. The statistical analyses will be handled in a descriptive manner. Descriptive statistics (frequency table) and histogram will be used to summarize clinical outcomes related to IIC.

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials